CLINICAL TRIAL: NCT05288829
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of a Single Dose of ALXN1210 Administered Subcutaneously Compared to Intravenously in Healthy Subjects
Brief Title: A Study of a Single Subcutaneous Dose of ALXN1210 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ALXN1210-SC-101; 2016-001617-24 (EudraCT Number)
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Pharmacodynamics; ALXN1210; Safety; Immunogenicity
MeSH Terms: interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: This was a partially blinded study. During Cohorts 1a and 1b dosing, participants, study site medical/nursing staff, and other study site staff involved in the safety evaluations were blinded to study drug assignment. The pharmacy staff who prepared the SC injections and the research physician responsible for study drug administration was not blinded. In addition, a data manager responsible for masking some of the PK data was not blinded. Alexion staff were unblinded only on specific occasions (eg, to monitor that the SC injections were being prepared appropriately, to determine reportability of serious adverse events [AEs]), and refrained from sharing any information on study drug assignment with the study site staff. During Cohort 2, however, participants and study site staff were made aware of the treatment being administered.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ALXN1210 SC (Experimental): Participants received ALXN1210 SC.
  Interventions: Drug: ALXN1210 SC
- ALXN1210 IV (Experimental): Participants received ALXN1210 IV.
  Interventions: Drug: ALXN1210 IV
- Placebo SC (Placebo Comparator): Participants received placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN1210 SC — All doses of ALXN1210 SC were administered by four 100-milligram (mg) SC injections of 1 milliliter (mL) each in the abdominal area. All four 1-mL injections were administered over a 15-minute period with at least 15 minutes between the end of injection in 1 participant and the start of injection in the next participant.
  Other Names: Ravulizumab; Ultomiris
  Arms: ALXN1210 SC
Drug: ALXN1210 IV — All doses of ALXN1210 IV were administered by IV infusion, using IV sets with in-line filters, at a maximum rate of 333 mL/hour, excluding interruption for safety or technical reason. There were at least 15 minutes between the end-of-infusion/injection in 1 participant and the start-of infusion/injection in the next participant.
  Other Names: Ravulizumab; Ultomiris
  Arms: ALXN1210 IV
Drug: Placebo — All doses of placebo SC were administered by four 100-mg SC injections of 1 mL each in the abdominal area. All four 1-mL injections were administered over a 15-minute period with at least 15 minutes between the end of injection in 1 participant and the start of injection in the next participant.
  Arms: Placebo SC

SUMMARY:
This study evaluated the safety and tolerability of a single dose of ALXN1210 subcutaneous (SC) compared to ALXN1210 intravenous (IV) in healthy participants and to determine the absolute bioavailability of ALXN1210 SC.

DETAILED DESCRIPTION:
The participants were randomly assigned in a 2:1 ratio to Cohort 1a in a blinded fashion to receive either a single dose of ALXN1210 SC 400 mg or single dose of placebo SC. The Safety Review Committee (SRC) evaluated the first 48 hours of postdose clinical safety data for participants in Cohort 1a to determine if enrollment into Cohorts 1b or 2 could begin. Following the SRC review, participants were randomly assigned in a 2:1 ratio to either Cohort 1b or Cohort 2. Within Cohort 1b, participants were blinded and further randomly assigned in a 5:1 ratio to receive either a single dose of ALXN1210 SC 400 mg or a single dose of placebo SC, respectively. The participants in Cohort 2 received a single dose of ALXN1210 IV 400 mg in an open-label fashion. Safety, PK, PD, and immunogenicity assessments were performed on the follow-up period after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index from 18 through 29.9 kilogram (kg)/square meter, inclusive, and weight between 50 and 100 kg, inclusive.
* QT interval corrected using Fridericia's formula ≤ 450 milliseconds (msec) for males and ≤ 470 msec for females at Screening and prior to dosing on Day 1.
* Was willing and was able to give written informed consent and complied with the study visit schedule.
* Documented vaccination with tetravalent meningococcal conjugate vaccine at least 56 days and not more than 3 years prior to dosing. Documentation must have included a positive serum bactericidal antibody titer to confirm an immune response before study drug administration.
* Vaccination with serogroup B meningococcal vaccine at least 56 days prior to dosing on Day 1, with a booster administered at least 28 days prior to dosing on Day 1, with at least 28 days between the first and second injections.
* Female participants of childbearing potential, if heterosexually active, must use highly effective contraception.

Exclusion Criteria:

* Participants who were in intimate and prolonged contact with (defined as living under the same roof or providing personal care to) people younger than 2 years of age or older than 65 years of age, or who were either immunocompromised or had 1 of the following underlying medical conditions: anatomic or functional asplenia (including sickle cell disease); congenital complement, properdin, factor D, or primary antibody deficiencies; acquired complement deficiencies (for example, those receiving eculizumab); or human immunodeficiency virus (HIV).
* Participants who were one of the following: professionals exposed to environments of greater risk for meningococcal disease; research, industrial, and clinical laboratory personnel routinely exposed to Neisseria meningitidis; military personnel during recruit training (military personnel could have been at increased risk of meningococcal infection when accommodated in close quarters); daycare center workers; those living on a college or university campus; and those who planned to travel during the course of the study to or had travelled to endemic areas for meningococcal meningitis (for example, India, Sub-Saharan Africa, or pilgrimage to Saudi Arabia for Hajj) within the past 6 months.
* History of any Neisseria infection.
* History of unexplained, recurrent infection, or infection requiring treatment with systemic antibiotics within 90 days prior to dosing.
* Evidence of HIV infection (HIV-1 or HIV-2 antibody titer).
* Acute or chronic hepatitis B virus infection. Hepatitis B surface antigen (HBsAg) testing was required for all participants prior to enrollment. Participants with positive HBsAg were not enrolled. For participants with negative HBsAg, the following testing algorithm was required: If hepatitis B core antibody (HBcAb) was negative, the participant was eligible to enroll and If HBcAb was positive, the hepatitis B surface antibody (HBsAb) was tested. (If both HBcAb and HBsAb were positive, the participant was eligible to enroll and If HBcAb was positive and HBsAb was negative, the participant was not enrolled.)
* Acute or chronic hepatitis C virus infection (evidenced by antibody titer).
* Active systemic viral or fungal infection within 14 days prior to dosing.
* Positive or indeterminate QuantiFERON-TB test which indicated possible tuberculosis (TB) infection.
* History of latent or active TB or exposure to endemic areas within 8 weeks prior to the Screening visit.
* Female participants who are breastfeeding or are heterosexually active and unwilling to practice contraception and are not postmenopausal.
* Positive serum pregnancy test at Screening or on Day -1.
* Serum creatinine greater than the upper limit of normal (ULN) of the reference range of the testing laboratory at Screening or on Day -1.
* Alanine aminotransferase or aspartate aminotransferase > ULN of the reference range of the testing laboratory at Screening or > 1.5*ULN of the reference range of the testing laboratory on Day -1.
* Any of the following hematology results: hemoglobin < 130 grams (g)/liter for males and < 115 g/L for females, hematocrit < 0.37 L/L for males and < 0.33 L/L for females, white blood cell count < 3.0*10^3/microliter (μL), absolute neutrophil count < 2.0*10^3/μL, and platelet count < 150 or > 400*10^3/μL at Screening or on Day -1. Complete blood count clinical laboratory results that were considered clinically relevant and unacceptable by the Investigator at Day -1.
* History of complement deficiency or complement activity below the normal reference range as evaluated by complement alternative pathway enzyme-linked immunosorbent assay at Screening.
* History of malignancy with the exception of a nonmelanoma skin cancer or carcinoma in situ of the cervix that had been treated with no evidence of recurrence.
* Participation in a clinical study within 30 days before initiation of dosing on Day 1 or use of any experimental small-molecule therapy within 30 days prior to dosing on Day 1.
* Participation in more than 1 clinical study of a monoclonal antibody (mAb), or participation in a clinical study of a mAb within the 12 months prior to screening, during which the participants was exposed to the active study drug. Participants who participated in only 1 study of a mAb could have been considered for enrollment if they completed that study more than 12 months prior to screening.
* Prior exposure to ALXN1210.
* Major surgery or hospitalization within 90 days prior to dosing.
* History of allergy to excipients of ALXN1210 (for example, polysorbate 80).
* Documented history of allergy to penicillin or cephalosporin.
* History of significant allergic reaction (for example, anaphylaxis or angioedema) to any product (food, pharmaceutical, etc).
* Smoked > 10 cigarettes daily (former smokers could have been permitted to enroll at the Investigator's discretion).
* Positive urine drug toxicology screen at Screening or on Day -1.
* Donation of plasma within 7 days prior to dosing. Donation or loss (excluding volume drawn at Screening) of more than 50 mL of blood within 30 days prior to dosing or more than 499 mL of blood within 56 days prior to dosing.
* Clinical diagnosis of any autoimmune or rheumatologic disease (for example, systemic lupus erythematosus, and rheumatoid arthritis).
* Immunization with a live-attenuated vaccine 28 days prior to dosing or planned vaccination during the course of the study (except for the vaccination planned per protocol). Immunization with inactivated or recombinant influenza vaccine was permitted.
* Presence of fever (confirmed body temperature > 37.6°C) (for example, a fever associated with a symptomatic viral or bacterial infection) within 14 days prior to dosing.
* Participants with any medical history, conditions, or risks that, in the opinion of the Investigator, could have interfered with the participant's full participation in the study or compliance with the protocol, or could have posed any additional risk for the participant or confounded the assessment of the participant or the outcome of the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 161 screened participants, 42 were randomly assigned to receive study drug: Placebo subcutaneous (SC), ALXN1210 400 milligrams (mg) SC, or ALXN1210 400 mg intravenous (IV).
Groups:
- ALXN1210 400 mg SC: Participants received a single dose of ALXN1210 400 mg via SC infusion on Day 1. Participants were followed for 200 days.
- ALXN1210 400 mg IV: Participants received a single dose of ALXN1210 400 mg via IV infusion on Day 1. Participants were followed for 200 days.
- Placebo SC: Participants received a single dose of placebo matched to ALXN1210 400 mg via SC infusion on Day 1. Participants were followed for 200 days.
Period: Overall Study
Arm/Group | ALXN1210 400 mg SC | ALXN1210 400 mg IV | Placebo SC
Started | 24 | 12 | 6
Received At Least 1 Dose Of Study Drug | 24 | 12 | 6
Completed | 24 | 12 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all participants who received the protocol-defined, single dose of study drug (ALXN1210 IV, ALXN1210 SC, or placebo SC).
Groups:
- Total: Total of all reporting groups
Arm/Group | ALXN1210 400 mg SC | ALXN1210 400 mg IV | Placebo SC | Total
Number analyzed (Participants) | 24 | 12 | 6 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (7.73) | 33.2 (8.20) | 34.2 (6.46) | 35.0 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 2 | 14
  Male | 16 | 8 | 4 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 23 | 11 | 6 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Number of participants based on race.
  participants
    Asian | 2 | 2 | 1 | 5
    Black or African American | 5 | 0 | 1 | 6
    White | 17 | 10 | 2 | 29
    Other | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or procedure, whether or not considered related to the medicinal product or procedure, which occurred during the course of the clinical study. TEAEs were defined as AEs with a start date or time on or after the first dose of the study drug. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Day 200
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1210 400 mg SC | ALXN1210 400 mg IV | Placebo SC
Number analyzed (Participants) | 24 | 12 | 6
Participants | 19 | 11 | 5

2. Primary Outcome: Absolute Bioavailability of ALXN1210 SC
Description: The absolute bioavailability of ALXN1210 SC is reported as the area under the serum concentration versus time curve from time 0 extrapolated to infinity (AUCinf) geometric mean of the ALXN1210 SC group divided by the AUCinf geometric mean of the ALXN1210 IV group*100. Linear mixed model with fixed and random effects for the participant was used.
Time Frame: Predose , end of infusion (EOI); 30 minutes post EOI; 2, 4, and 8 hours post start of infusion; and from Day 2 up to Day 150
Population: The pharmacokinetic (PK) population consisted of all participants from the safety population who received either ALXN1210 SC or ALXN1210 IV and who had sufficient serum concentration data to enable the calculation of PK parameters. For this outcome measure, the N includes the participants from both the SC and IV groups.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of ratio
Groups:
- ALXN1210 400 mg SC/IV: Participants received single dose of ALXN1210 400 mg via SC or IV infusion on Day 1. Participants were followed up for 200 days.
Arm/Group | ALXN1210 400 mg SC/IV
Number analyzed (Participants) | 36
percentage of ratio | 60.4 [49.7 to 73.3]

3. Secondary Outcome: Percent Change From Baseline in Free Complement Protein C5 Concentration At Day 8
Description: Blood samples were collected to determine the percent change in free C5 serum concentration from baseline over time.
Time Frame: Baseline, Day 8
Population: The pharmacodynamic (PD) population consisted of all participants from the safety population who had sufficient total and free C5 concentration data and chicken red blood cells (cRBC) hemolysis data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 400 mg SC | ALXN1210 400 mg IV | Placebo SC
Number analyzed (Participants) | 24 | 12 | 6
percent change | -77.08 (24.481) | -98.81 (0.707) | 6.40 (13.397)

4. Secondary Outcome: Percent Change From Baseline In Chicken Red Blood Cell Hemolysis At Day 8
Description: Blood samples were collected to determine the percent change in cRBC from baseline over time.
Time Frame: Baseline, Day 8
Population: The PD population consisted of all participants from the safety population who had sufficient total and free C5 concentration data and cRBC hemolysis data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 400 mg SC | ALXN1210 400 mg IV | Placebo SC
Number analyzed (Participants) | 24 | 12 | 6
percent change | -29.49 (33.278) | -66.72 (33.553) | -11.14 (9.330)

5. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADAs) to ALXN1210
Description: Blood samples were collected to evaluate antibody response through development of ADAs. The number of participants who developed ADAs (ADA positive) to ALXN1210 were reported in this outcome measure.
Time Frame: Baseline up to Day 200
Population: The immunogenicity analysis population consisted of all participants who had a pre-dose and post-dose ADA sample collected. ADA was data collected for the ALXN1210 arms (SC, IV) only.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1210 400 mg SC | ALXN1210 400 mg IV
Number analyzed (Participants) | 24 | 12
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 200
Description: The safety population consisted of all participants who received the protocol-defined, single dose of study drug (ALXN1210 IV, ALXN1210 SC, or placebo SC).
Arm/Group | ALXN1210 400 mg SC | ALXN1210 400 mg IV | Placebo SC
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 19/24 | 11/12 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ALXN1210 400 mg SC (N=24) | ALXN1210 400 mg IV (N=12) | Placebo SC (N=6)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 3 (3) | 3 (3)
Migraine (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (13) | 7 (8) | 5 (7)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Balanitis candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/8 (0) | 0/4 (0) | 1/2 (1) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT05288829/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05288829/SAP_001.pdf